CLINICAL TRIAL: NCT03648606
Title: Improvement of the Early Management and Thermal Comfort of Premature Infants Under 32 Weeks of Amenorrhea Placed in a Closed Incubator: Comparison of the Use of the Incubator in Conventional "Air" vs. "Cutaneous" Regulation Mode .
Brief Title: Management and Thermal Comfort of Premature Infants Under 32 Weeks
Acronym: CTNNP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI10-PR-TOURNEUX-1
Record Dates: First submitted 2018-08-01; First posted 2018-08-27 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2018-08

CONDITIONS: Thermoregulation
Keywords: infant; thermoregulation; wakefulness episode

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: mesure of skin temperature — The infants are placed in a closed incubator to study the variability of the heart and respiratory frequencies according to the regulation of the incubator and to quantify the time spent outside. Data will be collected during the first 10 days of life of the preterm infant. Skin temperatures at six body sites (the abdomen, pectoral region, eye, hand, thigh and foot) were measured (using infrared thermography) during nocturnal polysomnography in 29 9-day-old preterm neonates (postmenstrual age:
  209 9 days). The investigators then determined whether the duration of the W episode depended upon the local skin temperatures measured at the start, during and end of the episode.

SUMMARY:
Sleep propensity was assessed in terms of the duration of a spontaneous episode of wakefulness (W). Skin temperatures at six body sites (the abdomen, pectoral region, eye, hand, thigh and foot) were measured (using infrared thermography) during nocturnal polysomnography in 29 9-day-old preterm neonates (postmenstrual age: 209 9 days). Te investigators then determined whether the duration of the W episode depended upon the local skin temperatures measured at the start, during and end of the episode.

DETAILED DESCRIPTION:
Although sleep is of paramount importance for preterm neonates, care of the latter in a neonatal intensive care unit does not favour sleep. Given that several studies in adults have described a 'vegetative preparedness to sleep' (in which distal skin vasodilation before lights-out promotes rapid sleep onset), the investigators looked at whether or not this process operates in preterm neonates. Sleep propensity was assessed in terms of the duration of a spontaneous episode of wakefulness (W). Skin temperatures at six body sites (the abdomen, pectoral region, eye, hand, thigh and foot) were measured (using infrared thermography) during nocturnal polysomnography in 29 9-day-old preterm neonates (postmenstrual age: 209 9 days).

ELIGIBILITY:
Inclusion Criteria:

* premature newborns 25 to 32 weeks of amenorrhea;
* arrival in the Neonatal Medicine Unit <12 hours of life;
* need for management in a closed incubator;
* availability of an incubator equipped with communication card.

Exclusion Criteria:

* premature newborns> 32 weeks of amenorrhea;
* arrival in the Neonatal Medicine unit after 12 hours of life;
* presence of malformation syndrome or serious heart disease;
* pathology requiring management within the first 10 days of life;
* Apgar score <5 at 10 minutes of life;
* need for initial management in an open incubator;
* unavailability of an incubator equipped with a communication card

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants less than 32 weeks of amenorrhea admitted to birth in the Neonatal Medicine Unit will be included after obtaining written parental consent. Data will be collected during the first 10 days of life of the preterm infant.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2010-06-04 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Mesure of the Thermal confort of preterm infants less than 32 weeks | 10 days
  The objective of this study is to evaluate the thermal confort (variability of the heart and respiratory frequencies) of preterm infant placed in a clmosed incubator to reduce the thermal stress of the very premature newborn (< 32 weeks of amenorrhea) during the first 10 days of life.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tourneux, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No